CLINICAL TRIAL: NCT03280212
Title: Tranexamic Acid in the Treatment of Residual Chronic Subdural Hematoma: A Single-centre, Observer-blinded, Randomized Controlled Trial.
Brief Title: Tranexamic Acid in the Treatment of Residual Chronic Subdural Hematoma
Acronym: TRACE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Michael Cusimano, Neurosurgeon, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0176-GAP
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Tranexamic acid; TXA
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid Arm (Experimental): Tranexamic Acid 500 milligrams (MG)
  Participants of the Tranexamic Acid (TXA) arm will receive the study drug, TXA. Participants of average body weight (60-100kg) will receive TXA according to a 500mg three times daily (TID) dose regimen. Weight deviations from this range will see dose adjustments as follows: participants <60kg will receive 500mg two times daily (BID), and participants >100kg will receive 1000mg BID.
  Interventions: Drug: Tranexamic Acid 500 MG
- Control Arm (No Intervention): No intervention
  Participants in the control arm will not receive any additional intervention, medication, or placebo, and will serve as a comparative arm for the experimental arm.

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Tranexamic Acid 500mg oral tablets.
  Other Names: TXA
  Arms: Tranexamic Acid Arm

SUMMARY:
Chronic subdural hematoma (CSDH) is a common disease after minor head trauma, especially in elderly patients. This medical condition is characterized by blood collection in the subdural space, which can result in severe neurological impairment. Current standard of care is the evacuation of the CSDH by means of different surgical approaches. Although clinical and surgical outcomes are satisfying in most cases, considerable morbidity and mortality as well as recurrence rates of 3-31% are frequently reported. Therefore a non-surgical approach for the treatment of CSDH would be desirable. Tranexamic acid (TXA), an antifibrinolytic drug has been shown to decrease hematoma volume in a small cohort of patients suffering from CSDH. The present study is designed to test the hypothesis that TXA can reduce the volume of CSDH. Volume measurements of residual CSDH after burr-hole surgery will be performed during study course to quantify treatment success. The trial is designed as a randomized controlled pilot study, where half of the patients will be assigned to daily intake of TXA, whereas the other half will receive medical treatment according to current practice without TXA prescription. The primary endpoint of the study is defined as volume change in milliliters (mL) after 4-8 weeks of treatment. Secondary endpoints are hematoma volume change at 8-12 weeks, the rate of patients with resolution of the CSDH after 4-8 weeks and 8-12 weeks days, as well as the rate of reoperation during study course due to hematoma extension and neurological deterioration. Additionally the neurological outcome and the drug compatibility will be estimated as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic subdural hematoma, and have a planned or have received a unilateral or bilateral burr-hole craniostomy or mini-craniotomy
* Written informed consent (patient, power of attorney or substitute decision maker)
* Competence to take study medication properly and regularly or access to care giver that is able to comply with accurate study medication administration

Exclusion Criteria:

* Hypersensitivity to TXA or any of the ingredients
* Pregnancy
* Irregular menstrual bleeding with unidentified cause
* Acquired colour vision disturbances
* Acute and chronic renal insufficiency indicated by glomerular filtration rate (GFR) ≤ 30 mL/min
* Hematuria, caused by diseases of renal parenchyma
* Current alcohol abuse (as indicated by an Alcohol Use Disorders Identification Test (AUDIT) score of 10 or higher) drug abuse, or recreational drug use
* Concomitant intake of hormonal contraceptives, factor IX complex concentrates, and anti-inhibitor coagulant concentrates (factor VII, activated factor IX)
* Active, history, or increased risk of thrombotic events (including deep vein thrombosis, pulmonary embolism, cerebral venous thrombosis, arterial thrombotic events), symptomatic carotid stenosis, myocardial infarction, acute coronary syndrome, coronary artery disease, or consumption coagulopathy within the past 2 years
* History of angioplasty with cardiac stent placement or mechanical heart valve
* Active or history of brain pathologies such as stroke (hemorrhagic and ischemic), subarachnoid hemorrhage, or malignant brain tumors (glioma, metastasis and others) as well as history of seizures within the past 2 years
* Contraindication to stopping full therapeutic doses of non-acetylsalicylic acid (ASA) antiplatelets, warfarin, rivaroxaban, apixaban, dabigatran, or other anticoagulant for 2 weeks after surgery
* Patients requiring immediate revision surgery (as defined by attending surgeon)
* Inability of oral drug intake or missing support to guarantee oral drug intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Chronic subdural hematoma volume change | 4-8 weeks, 8-12 weeks
  Change in hematoma volume in mL according to volume measurements made on CT scans comparing CT scan at 4-8 weeks to immediate post-operative CT scan.

SECONDARY OUTCOMES:
Neurological outcome | 4-8 weeks, 8-12 weeks
  An assessment of neurological outcome as measured by the National Institutes of Health Stroke Scale (NIHSS)
Quality of life | 4-8 weeks, 8-12 weeks
  Participants quality of life as measured on the Health Utilities Index (HUI).
Quality of life | 4-8 weeks, 8-12 weeks
  Participants quality of life as measured on the 36-item Short Form Health Survey (SF-36).
Occurrence of adverse events | 4-8 weeks, 8-12 weeks
  Safety of the TXA dose regimen by monitoring incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided